CLINICAL TRIAL: NCT02048293
Title: Pharmacodynamic Differences Between Branded and Unbranded Remifentanil Molecules Available in Colombia for Tracheal Intubation of Adult Patients, 2012-2013
Brief Title: Pharmacodynamic Differences Between Branded and Unbranded Remifentanil Molecules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Collaborators: Hospital de San Jose (Other)
Responsible Party: Principal Investigator, Luis Eduardo Reyes Ortiz, MD, Physician, Anesthesiologist, Intensive Care Specialist, Professor Fundación Universitaria de Ciencias de la Salud, Hospital de San José, Bogotá D.C., Fundación Universitaria de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 326-3847-22
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Pain
Keywords: remifentanil; propofol; pharmacodynamic; total intravenous anesthesia; orotracheal intubation; heart rate; mean arterial pressure; Cooper intubation condition score
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group O (Active Comparator): Remifentanyl innovative molecule = Ultiva®
  Interventions: Drug: Remifentanyl, Ultiva®; Drug: Fada Remifentanilo
- Group A (Active Comparator): Remifentanyl comparator A = Remifentanil Laboratorios Chalver de Colombia S.A.
  Interventions: Drug: Remifentanil Laboratorios Chalver de Colombia S.A.; Drug: Fada Remifentanilo
- Group B (Active Comparator): Remifentanyl comparator B = Fada Remifentanilo
  Interventions: Drug: Remifentanyl, Ultiva®; Drug: Remifentanil Laboratorios Chalver de Colombia S.A.

INTERVENTIONS:
Drug: Remifentanyl, Ultiva® — Anesthetic induction for orotracheal intubation. Group O
  Arms: Group B; Group O
Drug: Remifentanil Laboratorios Chalver de Colombia S.A. — Anesthetic induction for orotracheal intubation. Group A
  Arms: Group A; Group B
Drug: Fada Remifentanilo — Anesthetic induction for orotracheal intubation. Group B
  Arms: Group A; Group O

SUMMARY:
Unbranded drug molecules are produced after the patent of a given drug has expired. Unbranded molecules of Remifentanil have been marketed in Colombia, and several reports by anesthesiologist indicate that there are differences in the physiologic response of patients to these molecules. The investigators hypothesized that unbranded molecules of remifentanil require higher doses to obtain desired physiological responses as compared to the branded molecule.

DETAILED DESCRIPTION:
Introduction. Several remifentanil products are commercialized in Colombia while these have never been compared in a clinical setting.

Objective. The aim of this study was to investigate the pharmacodynamic profile of the innovative molecule of remifentanil (group O = Ultiva®) and two unbranded molecules (group A = Remifentanil Laboratorios Chalver de Colombia S.A. and group B = Fada Remifentanilo) registered in Colombia.

Methods. The investigators carried out a double-blind, randomized, controlled trial. The branded molecule of remifentanil (group O, n=29) was compared against the two unbranded molecules (group A, n=29; group B, n=32) during anesthetic induction and tracheal intubation in adult patients American Society of Anesthesiology Physical Status Classification = I without predictors for difficult airway. The target controlled infusion (TCI) doses evaluated were 6, 8 and 10 ng/ml with the Minto model. Induction was complemented with propofol 5 mg/ml (TCI) with the Schneider model and rocuronium 0.6 mg/kg. The primary outcome was defined as the difference in mean arterial pressure and heart rate pre-intubation (TCI equilibrium) and post-intubation (maximum measurement within 5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring orotracheal intubation
* 18-50 years old
* Body mass index <31 kg/m2
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Risk of difficult airway
* History of opioid use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Composite outcome of heart rate or mean arterial pressure difference before and after tracheal intubation | Average of 5 minutes
  Heart rate measured with EKG. Mean arterial pressure measured with automatic blood pressure cuff.

SECONDARY OUTCOMES:
Cooper intubation condition score | Measured during tracheal intubation, average of 30 seconds
  Jaw relaxation: 0 poor, 1 minimum, 2 moderate, 3 good. Vocal cords: 0 closed, 1 closing, 2 moving, 3 open. Intubation response: 0 severe cough, 1 mild cough, 2 mild diaphragmatic movement, 3 no response.
  Cooper score: Jaw relaxation + Vocal cords + Intubation response

CONTACTS AND LOCATIONS:
Overall Officials: luis e reyes, professor, Principal Investigator — fundacion universitaria de ciencias de la salud
Locations (1):
- Fundación Universitaria de Ciencias de la Salud, Hospital de San Jose, Bogota, Cundinamarca, Colombia

REFERENCES:
- [Background] Kwak HJ, Min SK, Kim DH, Kang M, Kim JY. Effect-site concentration of remifentanil for nasotracheal versus orotracheal intubation during target-controlled infusion of propofol. J Int Med Res. 2011;39(5):1816-23. doi: 10.1177/147323001103900524. PMID 22117982
- [Background] Lysakowski C, Dumont L, Pellegrini M, Clergue F, Tassonyi E. Effects of fentanyl, alfentanil, remifentanil and sufentanil on loss of consciousness and bispectral index during propofol induction of anaesthesia. Br J Anaesth. 2001 Apr;86(4):523-7. doi: 10.1093/bja/86.4.523. PMID 11573626
- [Background] Coskun D, Celebi H, Karaca G, Karabiyik L. Remifentanil versus fentanyl compared in a target-controlled infusion of propofol anesthesia: quality of anesthesia and recovery profile. J Anesth. 2010 Jun;24(3):373-9. doi: 10.1007/s00540-010-0898-1. Epub 2010 Mar 13. PMID 20229001